CLINICAL TRIAL: NCT04470817
Title: Post-Marketing Surveillance (Usage Results Study) of Azilsartan Medoxomil in the Treatment of Adult Patients With Essential Hypertension in South Korea
Brief Title: A Study for PMS of AZL-M in the Treatment of Adult Participants With Essential Hypertension in South Korea
Status: Completed | Type: Observational
Sponsor: Celltrion Pharm, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-491-4001; U1111-1252-3589 (Registry Identifier: WHO)
Record Dates: First submitted 2020-07-13; First posted 2020-07-14 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Essential Hypertension
Keywords: Drug Therapy
MeSH Terms: conditions — Essential Hypertension | interventions — azilsartan medoxomil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Essential Hypertension: Participants diagnosed with essential hypertension and whom have been prescribed azilsartan medoxomil as a monotherapy or taken concomitantly with other anti-hypertension therapies in a routine clinical practical setting, will be observed prospectively over a period of 6 years.
  Interventions: Drug: Azilsartan Medoxomil

INTERVENTIONS:
Drug: Azilsartan Medoxomil — Azilsartan Medoxomil

SUMMARY:
The purpose of this study is to evaluate the safety by determining the incidence rates of all adverse events (AEs) including serious adverse events (SAEs)/serious adverse drug reactions (ADRs), unexpected AEs and ADRs that are not reflected on the precaution in the use, ADRs already known, non-serious ADRs and other safety related information (laboratory values changes, etc).

DETAILED DESCRIPTION:
This is a long-term prospective, observational post-marketing surveillance study of azilsartan medoxomil in participants with essential hypertension. This study will assess the safety and effectiveness of azilsartan medoxomil prescribed as a monotherapy or taken concomitantly with other anti-hypertension therapies in real-world clinical practice settings.

The study will enroll approximately 3000 participants. The data will be prospectively collected, at the centers from medical files and recorded into electronic case report forms (e-CRFs). All the participants will be assigned to a single observational cohort:

* Participants With Essential Hypertension

The multi-center study will be conducted in South Korea. Data collection will be based on routinely scheduled and emergency visits over the surveillance period, scheduled at Visit 1 (Baseline), Visit 2 (6 Weeks), Visit 3 (3 Months or more less than 6 Months) and Visit 4 (6 Months or more [Month 9]). The overall duration of the study will be approximately 6 years. All participants will be followed up for 9 months after drug administration.

ELIGIBILITY:
Inclusion Criteria:

1. With Essential Hypertension.

   * Newly diagnosed with essential hypertension or who have no long-term history of hypertension medication after diagnosis (The participant has a SBP or DBP >=140 or 90 mmHG, respectively).
   * Receiving treatment with other hypertension medications.
2. Newly prescribed and initiates azilsartan medoxomil for the treatment of hypertension, as a monotherapy or taken concomitantly with other anti-hypertension therapies.

Exclusion Criteria:

1. Treated with azilsartan medoxomil outside of the locally approved label in South Korea.
2. With known hypersensitivity or presence of any contraindication to azilsartan medoxomil.
3. Use of aliskiren in combination with azilsartan medoxomil in participants with diabetes or with moderate to severe renal impairment (glomerular filtration rate [GFR ] < 60 milliliter per minute [mL/min]/1.73 m^2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with essential hypertension and whom have been prescribed azilsartan medoxomil as a monotherapy or taken concomitantly with other anti-hypertension therapies in a routine clinical practical setting.
Sampling Method: Non-Probability Sample
Enrollment: 3438 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Experience at Least one AE and SAE | Baseline up to Month 9

SECONDARY OUTCOMES:
Change From Baseline in Blood Pressure Including Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) | Baseline up to Month 9
  Blood pressure (SBP and DBP) will be measured in millimeter of mercury (mmHg).
Percentage of Participants who Achieve Clinic DBP Less Than (<) 90 mmHg and/or Reduction of Greater Than or Equal to (>=) 10 mmHg | Baseline up to Month 9
Percentage of Participants who Achieve Clinic SBP <140 mmHg and/or reduction of >=20 mmHg | Baseline up to Month 9
Percentage of Participants who Achieve Both Clinic DBP <90 mmHg and/or Reduction of >=10 mmHg and Clinic SBP <140 mmHg and/or Reduction of >=20 mmHg | Baseline up to Month 9
Change From Baseline in Serum Creatinine Level, Serum Uric Acid Level and Serum Lipid Profile | Baseline up to Month 9
  Serum creatinine level, serum uric acid level, and serum lipid profile will be measured in milligram per deciliter (mg/dL).
Change From Baseline in Blood Potassium Level | Baseline up to Month 9
  Blood potassium level will be measured in millimole per liter (mmol/L).
Change From Baseline in Blood Sodium Profiles | Baseline up to Month 9
  Blood sodium profiles will be measured in milliequivalent per liter (mEq/L).
Final Effectiveness Rate as Assessed by the Investigator | Baseline up to Month 9
  Effectiveness rate: percentage of participants who achieved effectiveness over total number of assessable effectiveness analysis population, and is calculated as number of effective participants/total number of participants in group, multiplied by 100. Final effectiveness will be assessed based on: Improved (symptoms have improved or it is considered to have had a maintenance effect); Unchanged (no significant change from pre-administration, not considered to have had a maintenance effect); Worsened (symptoms have worsened compared to pre-administration); Unassessable (unable to assess due to grounds such as missing effectiveness variables, follow up loss, etc.). Maintenance effect: cases where the likelihood of worsened symptoms is high with discontinuation of medication, or equivalent effect to existing drugs is sustained when substituted with existing drugs. Effectiveness rate is determined by classifying 'Improved' as "Effective" and 'Unchanged' and 'Worsened' as "Ineffective".

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Celltrion Pharm, Inc.
Locations (1):
- Myongji Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.